CLINICAL TRIAL: NCT06066905
Title: A Study of Chidamide With AZA in MRD Positive AML After Transplant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Shenzhen Chipscreen Biosciences Co.Ltd (Unknown)
Responsible Party: Principal Investigator, WENG Jian yu, professor, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chidaza101
Record Dates: First submitted 2023-09-19; First posted 2023-10-04 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: AML, Adult; Minimal Residual Disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chidamide and azacitidine (Experimental)
  Interventions: Drug: chidamide and azacitidine

INTERVENTIONS:
Drug: chidamide and azacitidine — chidamide：10mg orally,day 1 to day 6 every week, Take it for two weeks, rest for two weeks,so 28 days for a circle, 12 circles totally.
  azacitidine:50mg,subcutaneous injection,day 1 to day 5 every week, 28 days for a circle, 6 circles totally.

SUMMARY:
acute myeloid leukemia (AML) is a malignant tumor of the hematopoietic system with high heterogeneity in cytogenetics and molecular biology.Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is still the primary treatment option for patients with AML and the most effective method for radical treatment of AML.Despite considerable progress in allo-HSCT over the past decade, 30%-40% of patients still relapse, and post-transplant relapse remains the leading cause of death in patients with AML.

DETAILED DESCRIPTION:
Investigators proposed Chidamide combined with azacitidine as the prospective treatment for MRD-positive AML patients before and after transplantation, hoping to reduce the recurrence rate of transplantation and improve the transplantation effect. The efficacy and safety of the method will be verified by this clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with AML (diagnostic criteria refer to WHO2016 criteria, except M3) can detect small residual lesions (MRD) positive after allogeneic hematopoietic stem cell transplantation (allo-HSCT);
2. ≥18 years old;
3. ECOG≤3;
4. lifespan≥3 months;
5. Take contraceptive measures;
6. Sign informed consent.

Exclusion Criteria:

1. Allergic to the study drug;
2. A gastrointestinal condition that prevents oral medication;
3. active infection;
4. Dysfunction of vital organs;
5. other malignancies;
6. HIV infection;
7. HBV or HCV;
8. The QT interval is prolonged;
9. Pregnant or lactating women;
10. Is participating in other clinical studies;
11. The researchers did not consider it appropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-26 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
the rate of RFS in 6 months | 6 months
  relapse-free survival

SECONDARY OUTCOMES:
the rate of MRD turn negative in 6 months | 6 months
  minimal residual disease turn negative
the time length of MRD negative | 24 months
  minimal residual disease negative
the 1 year/2 year RFS | 24 months
  relapse-free survival
the 1 year/2 year OS | 24 months
  overall survival
the rate of GVHD | 24 months
  graft-versus-host disease
Incidence of Treatment-Emergent Adverse Events | 24 months
  Grade 1 to Grade 4 ,according to Common Terminology Criteria for Adverse Events, versions 5.0

OTHER OUTCOMES:
T cell receptor excision circles (TRECs) level before and after treatment | 24 months
  T cell receptor excision circles (TRECs) are released upon rearrangement of the T cell receptor.
the rate of MRD turn negative in molecular genetic abnormality subtype | 24 months
  minimal residual disease

CONTACTS AND LOCATIONS:
Overall Officials: WENG jian yu, M.D., Principal Investigator — Department of Hematology, Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No